CLINICAL TRIAL: NCT05170048
Title: A Phase 2, Parallel, Randomized, Open-label, Controlled Study of EG-301 150 mg Daily in Patients With Nonfocal Geographic Atrophy Secondary to Dry-AMD
Brief Title: Study to Evaluate Safety and Efficacy of EG-301 in Patients With Nonfocal Geographic Atrophy Secondary to Dry-AMD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Evergreen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EG-301-2.1
Record Dates: First submitted 2021-12-10; First posted 2021-12-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Non-Exudative (Dry) Age-related Macular Degeneration (dAMD)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Arm: AREDS2 supplements (SOC) (Active Comparator): All patients assigned to this Control Group will receive standard of care to include AREDS2 supplements daily throughout the study.
  Interventions: Dietary Supplement: AREDS2 supplements
- Experomental Arm: AREDS2 supplements (SOC) plus EG-301 (Experimental): Patients assigned to the Experimental Group will receive a standard of care equivalent to that of the Control Group plus EG-DPMP-01 (150 mg daily, given at bedtime with a light snack).
  Interventions: Drug: EG-301; Dietary Supplement: AREDS2 supplements

INTERVENTIONS:
Drug: EG-301 — The investigation drug, EG-301 Tablets 150mg, is for oral use.
  Arms: Experomental Arm: AREDS2 supplements (SOC) plus EG-301
Dietary Supplement: AREDS2 supplements — AREDS2 supplement is the stand of care

SUMMARY:
This is a parallel, randomized, open-label, controlled study to evaluate the efficacy and safety of oral EG-301 in patients with intermediate non-exudative (dry) age-related macular degeneration (dAMD).

Ninety patients will be randomly allocated in a 2:1 ratio to one of two treatment arms for at least 6 months duration. The two treatment arms are:

1. AREDS2 supplements (Control Group, N=30)
2. AREDS2 supplements plus EG-DPMP-01 150 mg daily (Experimental Group, N=60)

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female patients, 50 to 75 years of age at screening visit
2. Subject has signed the Informed Consent form
3. Subjects with intermediate nonfocal geographic atrophy secondary to Non-Exudative (dry) AMD having ETDRS BCVA between 35 and 80 letters read (equivalent to 20/25 - 20/200 on Snellen Chart) with the level of vision caused by the non-exudative AMD and no other factor/s
4. Subjects with symptomatic decrease in visual acuity in the last 12 months
5. Subjects with confirmed diagnosis of geographic atrophy (GA) secondary to dAMD in the study eye* as evidenced by the following characteristics:

   * Non-center involving GA lesions that reside completely within the FAF imaging field (field 2, 30 degree image centered on the fovea)
   * Total GA area is ≥2.5 and ≤ 17.5 mm2 (1 and 7 disk areas [DA])
   * If GA is multifocal, at least one focal lesion must be >1.25 mm2 (0.5 DA)
   * Combination of areas of RPE disturbances described as a pattern of hyper or hypo-pigmentation in the junctional zone of GA. Absence of hyper-autofluorescence is exclusionary
6. Subjects with evidence of reasonably well-preserved areas of RPE by clinical examination and well-defined RPE and outer segment ellipsoid line by OCT examination in the central 1 mm of the macula as confirmed by the central reading center. More specifically, reasonably well- preserved central 1 mm of the macula means:

   * The RPE and outer retinal layers throughout the central 1 mm are intact
   * No signs of NVAMD such as intraretinal or sub retinal fluid, or sub retinal hyper-reflective material
   * No serous pigment epithelium detachments >100 microns in height
   * Sufficiently clear ocular media, adequate pupillary dilation, fixation to permit quality fundus imaging, and able to cooperate sufficiently for adequate ophthalmic visual function testing and anatomic assessment

Key Exclusion Criteria:

1. Females who are pregnant, nursing, planning a pregnancy during the study or who are of childbearing potential not using a reliable method of contraception and/or not willing to maintain a reliable method of contraception during their participation in the study. Women of childbearing potential with a positive urine pregnancy test administered at baseline are not eligible to receive study drug
2. Prior cataract surgery is allowed up to 90 days before the baseline visit, but refractive surgery in either eye may not be conducted during the study.
3. Subject with exudative AMD or choroidal neovascularization (CNV), including any evidence of retinal pigment epithelium rips, detachments or evidence of neovascularization anywhere in either eye based on SD-OCT imaging and/or fluorescein angiography as assessed by the Reading Center
4. Subjects who had anti-VEGF IVT in either eye in the past 90 days
5. Subjects who have received any drug or herbal medicine known to inhibit CYP2D6 enzyme activity prior to the first dose of the investigational drug (the patient can be enrolled if the washout period is ≥5 half-lives of the CYP2D6 inhibitor), or subjects who need to continue receiving these medications during the study period. (Refer to Appendix 1 for a list of CYP2D6 inhibitors)
6. Subjects with moderate or severe renal impairment as indicated by an estimated glomerular filtration rate (eGFR) <60 mL/min, calculated by using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events Assessment using CTCAE v5.0 | Evaluation in 26 weeks treatment period, and 4 weeks safety follow up period.
  Number of Participants With Treatment-Related Adverse Events as Assessed by NCI CTCAE v5.0, toxicities will be characterized in terms including seriousness, causality, toxicity grading, and action taken with regard to trial treatment.
GA lesion size change | From baseline to Week 26 treatment period
  The mean change in GA lesion size as measured by a) fundus autofluorescence (FAF) by an independent central reading center (CRC), and b) SD-OCT
Overall retinal sensitivity | From baseline to Week 26 treatment period
  Change in overall retinal sensitivity as measured by microperimetry using macular integrity assessment (MAIA)
BCVA in number of letters | From baseline to Week 26 treatment period, and 4 weeks safety follow up period.
  The mean change in BCVA in the number of letters as assessed by the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol
Low luminance visual acuity (LLVA) | From baseline to Week 26 treatment period
  The mean change in low luminance visual acuity (LLVA) in number of letters as assessed by the ETDRS protocol
Binocular reading speed | From baseline to Week 26 treatment period
  Binocular reading speed as assessed by the Minnesota Low-Vision Reading Test (MNRead) Charts
Binocular critical print size | From baseline to Week 26 treatment period
  Binocular critical print size as assessed by the Minnesota Low-Vision Reading Test (MNRead) Charts
NEI-VFQ score | From baseline to Week 26 treatment period
  Change in NEI-VFQ score

SECONDARY OUTCOMES:
Plasma levels of bioactive lipids | From baseline to Week 26 treatment period
  Changes in plasma levels of bioactive lipids, including sphingolipids, ceramides, and lysophosphatidic acids
Plasma levels of beclin-1 levels | From baseline to Week 26 treatment period
  Changes in plasma levels of beclin-1 levels as measured by the enzyme-linked immunosorbent assay (ELISA) method with a human beclin-1 ELISA kit
Complement factor levels | From baseline to Week 26 treatment period
  Changes in complement factor levels, including plasma concentrations of activation products C3d, Ba, C3a, C5a, and SC5b-9.